CLINICAL TRIAL: NCT01686048
Title: The Significance of Ambrosia in Allergic Rhinitis and Asthma in Israel
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Arnon Goldberg, Head, Allergy and Clinical Immunology Unit, Meir Medical Center
Other Study IDs: Ambrosia
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Allergic Rhinitis; Asthma; Allergic Conjunctivitis; Atopic Dermatitis
MeSH Terms: conditions — Rhinitis, Allergic; Asthma; Conjunctivitis, Allergic; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Ambrosia is known for its allergenicity in the USA causing hay fever and asthma. Israel has always been considered "clean" of Ambrosia but over the past years growth of Ambrosia plants has been detected in several locations in Israel.

In the proposed study, patients referred for routine allergic evaluation will also be skin tested with Ambrosia allergens, in addition to their regular prick skin tests with all other airborne allergens.

ELIGIBILITY:
Inclusion Criteria:

* Patients with allergic rhinitis, asthma, allergic conjunctivitis or atopic dermatitis who undergo prick skin tests with airborne allergens

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients refered for allergic evaluation
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Arnon Goldberg, M.D., Allergy and Clinical Immunology Unit, Meir Medical Center, Kfar Saba, Israel